CLINICAL TRIAL: NCT00786084
Title: Randomized Prospective Controlled Trial of Paraesophageal Hernia Repair With Small Intestine Submucosa (SIS)
Brief Title: Study of Paraesophageal Hernia Repair With Small Intestine Submucosa
Acronym: PEH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Cook Biotech Incorporated (Industry); Washington University School of Medicine (Other); Oregon Health and Science University (Other); The Oregon Clinic (Other)
Responsible Party: Brant Oelschlager, MD/Associate Professor, University of Washington
Other Study IDs: 21065-A
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Hiatal Hernia; Paraesophageal Hernia
Keywords: Hiatal hernia; PEH; paraesophageal hernia; synthetic mesh; small intestine submucosa
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — None retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Phase I patients who had a paraesophageal hernia repair with synthetic mesh.
- 2: Phase I patients who had a paraesophageal hernia repair with small intestine submucosa mesh.

SUMMARY:
In 2006 this research group reported their initial findings of a multi-center prospective trial comparing primary repair and primary repair buttressed with a biologic mesh made from porcine small intestinal submucosa (SIS). We were able to accrue 108 patients from 7/2002-3/2005 and followed each patient over 6 months and performed an UGI to check the durability of the repair and rule out a recurrence. The results suggested a significant benefit for the use of SIS mesh in the short-term, with the primary group having a 26% recurrence rate and the mesh group a 9% recurrence rate.

While these results are encouraging, it is important to know what is the durability and the longer term benefits of the use of SIS mesh. For this reason we propose a follow-up of the original study patients with the same outcome measures (symptom questionnaire, SF-36, and UGI). This should give us a very good idea about the long-term success of laparoscopic PEH repair with primary and SIS mesh.

DETAILED DESCRIPTION:
Traditionally paraesophageal hernias were repaired by thoracotomy or laparotomy with morbidity around 20% and mortality of 2%.1,2 The advent and later popularization of antireflux operations via the minimally invasive approach led to the development of a similar (laparoscopic) approach to the treatment of paraesophageal hernia. This approach called for the excision of the sac, a thorough esophageal mobilization, primary closure of the hiatus and a Nissen fundoplication. 3,4 Laparoscopy appears to have some of the benefits of thoracotomy (the hiatus can be accessed easier, the esophagus can be dissected under direct vision and high mobilization of the esophagus is possible) and some of the advantages of the laparotomy (less morbidity, no need to collapse the lung, no need for postoperative chest tube). In fact, most PEH are currently repaired via a laparoscopic approach.

Hashemi et al in 2000 reported that patients who had had a repair of a paraesophageal hernia via the laparoscopic approach had a higher recurrence rate when compared to those operated on via thoracotomy and laparotomy.5 The only other study comparing open and laparoscopic repair revealed a higher incidence of recurrence in the open repair group (8% vs. 0%),6 but was also based solely on symptoms. Case series of LPEHR which evaluate recurrent hiatal hernia by x-ray or endoscopy have found the recurrence rate to be between 12-42%,3,5,7 suggesting significant room for improvement.

It is not surprising that primary repair of the paraesophageal hiatal hernia by suturing the pillars of the diaphragm together under tension is at significant risk for disruption. With the development and wide application of mesh materials for tension-free repair of inguinal and ventral hernias, many surgeons have applied the technique of tension-free closure with a mesh to the hiatal hernia. Two randomized trials have demonstrated a significant reduction in recurrence rates by using synthetic mesh in large hiatal hernia repairs.8,9 However, there are potential problems introduced by using synthetic mesh at the dynamic hiatus such as mesh erosion, ulceration, stricture, and dysphagia.9,10,11 Recently, a number of biomaterials have been developed for hernia repair. The idea behind them is that a biologic scaffold, usually containing extracellular collagen, serves as a temporary matrix, thus strengthening a natural hernia closure.12,13 One such mesh is derived from porcine small intestinal submucosa (SIS) (Cook Surgical Indianapolis, IN). A pilot study using SIS for PEH repair suggested that is was safe and possibly effective in reducing recurrence.14 We then organized and carried out a multi-center randomized trial comparing primary repair of the crura and buttressing a primary repair with SIS mesh during laparoscopic PEH repair. The results at 6 months after operation demonstrated a nearly 3-fold reduction in the recurrence rate with the use of mesh (26% to 9%).15 Furthermore, there were no mesh related complications such as dysphagia, infection, or erosion. These results have been met with tempered enthusiasm in the surgical community. The only question in many surgeon's minds is whether buttressed repair of the hiatus is durable. To answer this question we need to complete longer term follow-up in these patients.

The aim of this study is to determine if the use of SIS to reinforce the closure of the hiatus in patients with paraesophageal hernias results in a lower recurrence rate at 2.5-5 years after operation, and results in improved outcomes, without an increase in the complication rate.

ELIGIBILITY:
Inclusion criteria:

* Prior enrollment in Phase I study.

Exclusion criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prior enrollment in the Phase I study.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To determine the medium/long-term effect of SIS on recurrence rates after laparoscopic PEH repair. | One year

SECONDARY OUTCOMES:
Determine the objective durability of laparoscopic PEH repair with and without SIS | One year
Determine medium/long-term symptomatic outcomes of laparoscopic PEH repair with and without SIS | One year
Determine medium/long-term QOL outcomes of laparoscopic PEH repair with and without SIS | One year
Determine the incidence of long-term complications of SIS mesh for PEH repair (i.e. dysphagia, erosion, infection) | One year
Determine the durability of laparoscopic paraesophageal hernia repair with regard to a) anatomic recurrence b) symptom control | One year

CONTACTS AND LOCATIONS:
Overall Officials: Brant K Oelschlager, MD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - The Oregon Clinic, PC, Portland, Oregon
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Oelschlager BK, Pellegrini CA, Hunter J, Soper N, Brunt M, Sheppard B, Jobe B, Polissar N, Mitsumori L, Nelson J, Swanstrom L. Biologic prosthesis reduces recurrence after laparoscopic paraesophageal hernia repair: a multicenter, prospective, randomized trial. Ann Surg. 2006 Oct;244(4):481-90. doi: 10.1097/01.sla.0000237759.42831.03. PMID 16998356